CLINICAL TRIAL: NCT00329784
Title: Induction of Tolerance Through Early Introduction of Peanut in High-Risk Children (ITN032AD)
Brief Title: Promoting Tolerance to Peanut in High-Risk Children
Acronym: LEAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN032AD
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Eczema; Egg Allergy; Food Allergy
Keywords: peanut allergy; egg allergy; eczema; peanut; allergy; allergies; allergic reaction; anaphylaxis; infants; children
MeSH Terms: conditions — Eczema; Egg Hypersensitivity; Food Hypersensitivity; Peanut Hypersensitivity; Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut Consumption Group (Experimental): Participants on this arm will consume peanut protein.
  Interventions: Biological: Peanut Consumption Group
- Peanut Avoidance Group (No Intervention): Participants on this arm will avoid peanut as per United Kingdom (UK) public health recommendations.

INTERVENTIONS:
Biological: Peanut Consumption Group — Peanut-containing snack. Children are to consume 2 g of peanut protein in three servings per week (total of 6 g) over 3 servings.
  Other Names: Bamba
  Arms: Peanut Consumption Group

SUMMARY:
This study will evaluate whether early exposure to peanuts promotes tolerance and provides protection from developing peanut allergy in children who are allergic to eggs or who have severe eczema.

This study has been continued into the ITN049AD (LEAP-On) Study (NCT01366846).

DETAILED DESCRIPTION:
Allergic reactions to peanuts are potentially life-threatening and, in some children, can result from ingestion of only trace quantities of peanuts. At highest risk are children with eczema or who are allergic to eggs; these children have a 20% chance of developing peanut allergy by the age of five. The majority of children allergic to peanuts have their first reaction between the ages of 14 and 24 months, often at the time of their first exposure to peanut. Currently, there is no cure for peanut allergy.

Peanut allergy has become an increasingly common problem in early childhood in the United States and the United Kingdom. Despite current public health guidelines in both countries recommending the avoidance of peanut consumption in the first years of life, the proportion of children with peanut allergy doubled in these countries over the period from 1998 to 2003. In contrast, peanuts are commonly consumed by infants in relatively high amounts in Africa, Southeast Asia and Israel, yet the rate of peanut allergy is quite low and does not appear to be increasing. Peanut consumption by infants in these parts of the world may actually protect children from developing peanut allergy by promoting oral tolerance to peanuts.

Participants in this study will be randomly assigned to either follow a peanut consumption regimen or a strict peanut avoidance regimen. Those assigned to the peanut consumption group will be asked to consume an age-appropriate snack three times a week for the duration of the study and will be monitored closely during their first introduction to peanut.

Those assigned to the peanut avoidance group will be asked to avoid ingestion of peanut for the first three years of life. A physical exam, allergy testing, and other immune system tests requiring blood collection will occur at Years 1, 3, and 5 following study entry. During the study, parents will maintain regular contact with study dietitians.

ELIGIBILITY:
Inclusion Criteria:

* Able to consume solid food
* Allergy to eggs and/or severe eczema
* Informed consent obtained from parent or guardian.

Exclusion Criteria:

* Clinically significant chronic illness. Participants with eczema or recurrent wheeze are not excluded.
* Positive skin prick test for peanut allergen with a wheel diameter greater than 4 mm in the presence of a negative saline control
* Previous or current consumption of peanut protein that exceeds 0.2 g of peanut protein on at least one occasion or 0.5 g over a single week
* Investigator-suspected allergy to peanut protein
* Investigator-suspected allergy to peanut protein in care provider or current household member.
* Diagnosis of persistent asthma
* ALT (SGPT) or bilirubin greater than 2 times the upper limit of age-related normal value
* BUN or creatinine greater than 1.25 times the upper limit of age-related normal value
* Platelet count less than 100,000/mL, hemoglobin less than 9 g/dL, or investigator-suspected immunocompromise
* Unwillingness or inability to comply with study requirements and procedures

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 640 (Actual)
Dates: Start 2006-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Lack, MD, Principal Investigator — Imperial College, St. Mary's Hospital
Locations (1):
- Evelina Children's Hospital, Guy's & St Thomas' NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in: 1.)ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools that are available to researchers who register online; and 2.)TrialShare, a clinical trials research portal of the Immune Tolerance Network (ITN).
Time Frame: Data sets et al of the manuscript are available to the public in TrialShare.
Access Criteria: The study ID in TrialShare is LEAP ITN032AD. Access is available to the public.
URL: https://www.itntrialshare.org/project/Studies/ITN032ADPUBLIC/Study%20Data/begin.view?pageId=study.DATA_ANALYSIS

REFERENCES:
- [Background] Palmer K, Burks W. Current developments in peanut allergy. Curr Opin Allergy Clin Immunol. 2006 Jun;6(3):202-6. doi: 10.1097/01.all.0000225161.60274.31. PMID 16670515
- [Background] Santos AF, Du Toit G, Lack G. Is the use of epinephrine a good marker of severity of allergic reactions during oral food challenges? J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):429-30. doi: 10.1016/j.jaip.2014.12.009. No abstract available. PMID 25956314
- [Background] Du Toit G, Sayre PH, Roberts G, Sever ML, Lawson K, Bahnson HT, Brough HA, Santos AF, Harris KM, Radulovic S, Basting M, Turcanu V, Plaut M, Lack G; Immune Tolerance Network LEAP-On Study Team. Effect of Avoidance on Peanut Allergy after Early Peanut Consumption. N Engl J Med. 2016 Apr 14;374(15):1435-43. doi: 10.1056/NEJMoa1514209. Epub 2016 Mar 4. PMID 26942922
- [Result] Du Toit G, Roberts G, Sayre PH, Bahnson HT, Radulovic S, Santos AF, Brough HA, Phippard D, Basting M, Feeney M, Turcanu V, Sever ML, Gomez Lorenzo M, Plaut M, Lack G; LEAP Study Team. Randomized trial of peanut consumption in infants at risk for peanut allergy. N Engl J Med. 2015 Feb 26;372(9):803-13. doi: 10.1056/NEJMoa1414850. Epub 2015 Feb 23. PMID 25705822
- [Result] Gruchalla RS, Sampson HA. Preventing peanut allergy through early consumption--ready for prime time? N Engl J Med. 2015 Feb 26;372(9):875-7. doi: 10.1056/NEJMe1500186. Epub 2015 Feb 23. No abstract available. PMID 25705823
- [Result] Du Toit G, Roberts G, Sayre PH, Plaut M, Bahnson HT, Mitchell H, Radulovic S, Chan S, Fox A, Turcanu V, Lack G; Learning Early About Peanut Allergy (LEAP) Study Team. Identifying infants at high risk of peanut allergy: the Learning Early About Peanut Allergy (LEAP) screening study. J Allergy Clin Immunol. 2013 Jan;131(1):135-43.e1-12. doi: 10.1016/j.jaci.2012.09.015. Epub 2012 Nov 19. PMID 23174658
- [Result] Feeney M, Du Toit G, Roberts G, Sayre PH, Lawson K, Bahnson HT, Sever ML, Radulovic S, Plaut M, Lack G; Immune Tolerance Network LEAP Study Team. Impact of peanut consumption in the LEAP Study: Feasibility, growth, and nutrition. J Allergy Clin Immunol. 2016 Oct;138(4):1108-1118. doi: 10.1016/j.jaci.2016.04.016. Epub 2016 Jun 10. PMID 27297994
- [Derived] Kanchan K, Cerosaletti K, Perry JA, DuToit G, Manohar M, Ling H, Paschall JE, Sanda S, Chinthrajah RS, Nepom GT, Nadeau KC, Jones SM, Lack G, Ruczinski I, Mathias RA. Genetic Determinants of Peanut-Specific IgG4 Levels in the Context of Sustained Oral Peanut Exposure in the LEAP Study. Immunology. 2026 Jan 30. doi: 10.1111/imm.70098. Online ahead of print. PMID 41615410
- [Derived] Roberts G, Bahnson HT, Du Toit G, O'Rourke C, Sever ML, Brittain E, Plaut M, Lack G. Defining the window of opportunity and target populations to prevent peanut allergy. J Allergy Clin Immunol. 2023 May;151(5):1329-1336. doi: 10.1016/j.jaci.2022.09.042. Epub 2022 Dec 12. PMID 36521802
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- See also: LEAP Study informational website — http://www.leapstudy.co.uk
- Available data/document: Individual Participant Data Set: SDY660 — https://immport.niaid.nih.gov/home — ImmPort study identifier is SDY660
- Available data/document: Study summary, -design, -adverse event(s), -demographics, -study files: SDY660 — https://immport.niaid.nih.gov/home — ImmPort study identifier is SDY660
- Available data/document: Individual Participant Data Set: LEAP (ITN032AD) — https://www.itntrialshare.org/project/Studies/ITN032ADNEJM/Study%20Data/begin.view?pageId=study.PARTICIPANTS — TrialShare study identifier is LEAP (ITN032AD)
- Available data/document: Overview, Date & Reports, Manuscripts et al.: LEAP (ITN032AD) — https://www.itntrialshare.org/project/Studies/ITN032ADNEJM/Study%20Data/begin.view? — TrialShare study identifier is LEAP (ITN032AD)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants between 4 and 11 months of age with pre-existing allergy to egg and/or severe eczema were recruited in the United Kingdom between December 2006 and May 2009.
Pre-assignment Details: Participants were stratified into cohorts based on a skin prick test for peanut allergen. Participants were either negative (no measureable wheal after test) or positive (a wheal measuring between 1 and 4 mm in diameter). Participants were then randomized into treatment groups.
Groups:
- Negative Stratum - Peanut Avoidance Group: Participants who had a negative response to a skin prick test for peanut allergen (no measurable wheal) and were then randomized to the peanut avoidance group. Participants were instructed to avoid exposure to peanut protein during study participation.
- Negative Stratum - Peanut Consumption Group: Participants who had a negative response to a skin prick test for peanut allergen (no measurable wheal) and were then randomized to the peanut consumption group. Participants were fed at least 2 g of peanut protein 3 times per week (a total of 6g). The preferred peanut source was Bamba (a peanut snack), although peanut butter was an acceptable substitute. After age 3, participants were allowed to eat whole peanuts.
- Positive Stratum - Peanut Avoidance Group: Participants who had a positive response to a skin prick test for peanut allergen (a wheal measuring between 1 and 4 mm) and were then randomized to the peanut avoidance group. Participants were instructed to avoid exposure to peanut protein during study participation.
- Positive Stratum - Peanut Consumption Group: Participants who had a positive response to a skin prick test for peanut allergen (a wheal measuring between 1 and 4 mm) and were then randomized to the peanut consumption group. Participants were fed at least 2 g of peanut protein 3 times per week (a total of 6g). The preferred peanut source was Bamba (a peanut snack), although peanut butter was an acceptable substitute. After age 3, participants were allowed to eat whole peanuts.
Period: Overall Study
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group
Started | 270 | 272 | 51 | 47
Completed | 265 | 267 | 51 | 47
Not Completed | 5 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group | Total
Number analyzed (Participants) | 270 | 272 | 51 | 47 | 640
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.7 (1.7) | 7.7 (1.8) | 8.4 (1.7) | 7.9 (1.6) | 7.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 124 | 17 | 19 | 256
  Male | 174 | 148 | 34 | 28 | 384
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 270 | 272 | 51 | 47 | 640
Severe Eczema [Count of Participants; unit: Participants] — Number of participants with severe eczema at baseline. Eczema is any type of dermatitis or inflammation of the skin. Severe eczema for this trial is based on three criteria. The first criterion was the parent or guardians' description of their child's eczema severity. The second criterion was the use of topical creams or ointments containing corticosteroids or calcineurin inhibitors. The third criterion will be a modified Scoring Atopic Dermatitis System (SCORAD). Infants with severe eczema are at a high risk of developing a peanut allergy
  Participants | 236 | 246 | 48 | 41 | 571
Age at Onset of Eczema [Mean (Standard Deviation); unit: Months] — Age in months at which eczema symptoms began. Eczema is any type of dermatitis or inflammation of the skin. Severe eczema for this trial is based on three criteria. The first criterion was the parent or guardians' description of their child's eczema severity. The second criterion was the use of topical creams or ointments containing corticosteroids or calcineurin inhibitors. The third criterion will be a modified Scoring Atopic Dermatitis System (SCORAD). Infants with severe eczema are at a high risk of developing a peanut allergy
  Months | 2.2 (1.7) | 2.3 (1.6) | 2.1 (1.6) | 2.4 (1.5) | 2.3 (1.6)
SCORAD [Mean (Standard Deviation); unit: units on a scale] — A modified Scoring Atopic Dermatitis System (SCORAD) was used to detect eczema in children who may not have had access to topical anti-inflammatory medications or whose parents cannot recall or report the severity of their child's eczema. Eczema is any type of dermatitis or inflammation of the skin. Atopic dermatitis is the most severe and chronic of all types of eczema. The range of the SCORAD is 0-103. Scores less than 15 indicate mild eczema, scores between 15 and 40 indicate moderate eczema, and scores greater than 40 indicate severe eczema.
  units on a scale | 35.0 (19.9) | 33.3 (18.4) | 33.7 (16.2) | 37.8 (18.6) | 34.4 (18.9)
Total IgE [Mean (Standard Deviation); unit: kUA/L] — Total Immunoglobulin E (IgE) includes the following potential allergens: peanut, hen's egg white, cow's milk, sesame, brazil nut, hazel nut, cashew, almond, walnut, house dust mite, cat dander, dog dander, timothy grass pollen, alternaria mold, and birch tree pollen. IgE is measured in a serum sample. Results <75 kUA/L suggests that the participant is not allergic to any of the potential allergens. A result >75 kUA/L suggests at least a mild clinical allergy. The higher the total IgE present in the serum sample, the more likely it is to be a presence of an allergy to at least one allergen
  kUA/L | 95.1 (321.8) | 76.4 (181.4) | 125.7 (174.8) | 306.4 (666.5) | 104.8 (307.9)
Peanut-specific IgE [Median (Inter-Quartile Range); unit: kUA/L] — Immunoglobulin E (IgE) is an antibody produced by the immune system. If you have an allergy, your immune system overreacts to an allergen by producing antibodies called IgE. These antibodies travel to cells that release chemicals, causing an allergic reaction. Peanut-specific IgE is measured in a serum sample following a peanut skin prick test. Results <0.35 kUA/L is considered low level allergic reaction to peanut. Results from >= 0.35 to <15 kUA/L are considered mid-level allergic reaction to peanut. Results >=15 kUA/L are considered high level allergic reaction to peanut.
  kUA/L | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.1] | 0.4 [0.1 to 3.0] | 1.3 [0.2 to 5.5] | 0.0 [0.0 to 0.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peanut Allergy at 60 Months of Age - by Skin Prick Test Stratum
Description: At 60 months of age, participants were given an oral food challenge Participants regarded as unlikely to be allergic to peanut received 5 g of peanut protein in a single dose. These participants were considered to have a peanut allergy if they experienced any type of reaction following consumption. A double-blind, placebo-controlled food challenge was offered to other participants with a total of 9.4 g of peanut protein administered in increments. These participants were considered to have a peanut allergy if at any point during the dose escalation procedure the participant had a reaction. Participants for whom data from the oral food challenge were either inconclusive or not available, a diagnostic algorithm based on clinical history, the results of a skin-prick test, and the values for peanut-specific IgE were used to determine whether or not a participant should be considered to have peanut allergy.
Time Frame: 60 months
Population: Intent-to-treat - all randomly assigned participants who were evaluable for peanut allergy at age 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group
Number analyzed (Participants) | 263 | 267 | 51 | 47
Participants | 36 | 5 | 18 | 5
Statistical Analysis 1: Comparison: Negative Stratum - Peanut Avoidance Group vs Negative Stratum - Peanut Consumption Group; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Positive Stratum - Peanut Avoidance Group vs Positive Stratum - Peanut Consumption Group; Test type: Superiority or Other; p = 0.004, Chi-squared

2. Primary Outcome: Number of Participants With Peanut Allergy at 60 Months of Age - Both Strata Combined
Description: as for outcome 1
Time Frame: 60 months
Population: Intent-to-treat - all randomly assigned participants who were evaluable for peanut allergy at age 60 months
Measure: Count of Participants; unit: Participants
Groups:
- Peanut Avoidance Group: Participants assigned to the peanut avoidance group were instructed to avoid exposure to peanut protein during study participation.
- Peanut Consumption Group: Participants assigned to the peanut consumption group were fed at least 2 g of peanut protein 3 times per week (a total of 6g). The preferred peanut source was Bamba (a peanut snack), although peanut butter was an acceptable substitute. After age 3, participants were allowed to eat whole peanuts.
Arm/Group | Peanut Avoidance Group | Peanut Consumption Group
Number analyzed (Participants) | 314 | 314
Participants | 54 | 10
Statistical Analysis 1: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Test type: Superiority or Other; p < 0.0001, Chi-squared

3. Secondary Outcome: SCORAD at 60 Months
Description: At 60 months of age, participants were assessed for eczema using a modified Scoring Atopic Dermatitis System (SCORAD). This measure was used to detect eczema in children who may not have had access to topical anti-inflammatory medications or whose parents cannot recall or report the severity of their child's eczema. Eczema is any type of dermatitis or inflammation of the skin. Atopic dermatitis is the most severe and chronic of all types of eczema. The range of the SCORAD is 0-103. A score of 0 indicates no eczema, scores between 0 and 15 indicate mild eczema, scores between 15 and 40 indicate moderate eczema, and scores greater than 40 indicate severe eczema.
Time Frame: 60 months
Population: Intent-to-treat with SCORAD data available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peanut Avoidance Group | Peanut Consumption Group
Number analyzed (Participants) | 316 | 312
units on a scale | 7.6 (11.6) | 6.6 (10.7)
Statistical Analysis 1: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Test type: Superiority or Other; p = 0.369, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Asthma at 60 Months
Description: At 60 months of age, participants were assessed for asthma. Participants were considered to have asthma if they had a history of cough, wheeze, or shortness of breath that (1) was responsive to therapy with bronchodilators on two or more occasions in the previous 24 months, (2) required one visit to a physician in the previous 24 months, or (3) occurred during the night, during early morning, or upon exercising in the intervals between exacerbations at any time in the previous 12 months.
Time Frame: 60 months
Population: Intent-to-treat with asthma data available
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Avoidance Group | Peanut Consumption Group
Number analyzed (Participants) | 316 | 314
Participants | 50 | 54
Statistical Analysis 1: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Test type: Superiority or Other; p = 0.642, Chi-squared

5. Secondary Outcome: Number of Participants With Rhinitis at 60 Months
Description: At 60 months of age, participants were assessed for rhinitis. Two types of rhinitis were assessed, perennial rhinoconjunctivitis and seasonal rhinoconjunctivitis. Participants were considered to have either type of rhinitis if they showed a sensitization to the allergen and clinical history of rhinoconjunctivitis symptoms experienced either when exposed to the relevant allergen (perennial) or during the relevant season (seasonal).
Time Frame: 60 months
Population: Intent-to-treat with rhinitis data available
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Avoidance Group | Peanut Consumption Group
Number analyzed (Participants) | 315 | 313
Participants
  Seasonal Rhinoconjunctivitis | 106 | 115
  Perennial Rhinoconjunctivitis | 134 | 132
Statistical Analysis 1: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Seasonal Rhinoconjunctivitis; Test type: Superiority or Other; p = 0.417, Chi-squared
Statistical Analysis 2: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Perennial Rhinoconjunctivitis; Test type: Superiority or Other; p = 0.926, Chi-squared

6. Secondary Outcome: Number of Participants With Specific Skin Prick Test Greater Than or Equal to 3mm
Description: At 60 months of age, participants were assessed for potential allergy to selected food allergens. Participants were considered to have a specific sensitivity if a skin prick containing the allergen produced a wheal size measuring greater than or equal to 3 mm.
Time Frame: 60 months
Population: Intent-to-treat with data available
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Avoidance Group | Peanut Consumption Group
Number analyzed (Participants) | 321 | 319
Participants
  Peanut Wheal: number analyzed (Participants) | 316 | 313
  Peanut Wheal | 71 | 30
  Egg Wheal: number analyzed (Participants) | 311 | 297
  Egg Wheal | 96 | 102
  Milk Wheal: number analyzed (Participants) | 308 | 298
  Milk Wheal | 28 | 25
  Sesame Wheal: number analyzed (Participants) | 305 | 287
  Sesame Wheal | 22 | 22
  Brazil nut Wheal: number analyzed (Participants) | 306 | 285
  Brazil nut Wheal | 29 | 26
  Hazel nut Wheal: number analyzed (Participants) | 306 | 284
  Hazel nut Wheal | 34 | 41
  Cashew Wheal: number analyzed (Participants) | 307 | 286
  Cashew Wheal | 42 | 59
  Walnut Wheal: number analyzed (Participants) | 306 | 283
  Walnut Wheal | 27 | 34
  Almond Wheal: number analyzed (Participants) | 305 | 283
  Almond Wheal | 42 | 50
Statistical Analysis 1: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Peanut Wheal; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Egg Wheal; Test type: Superiority or Other; p = 0.361, Chi-squared
Statistical Analysis 3: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Milk Wheal; Test type: Superiority or Other; p = 0.760, Chi-squared
Statistical Analysis 4: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Sesame Wheal; Test type: Superiority or Other; p = 0.834, Chi-squared
Statistical Analysis 5: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Brazil Nut Wheal; Test type: Superiority or Other; p = 0.882, Chi-squared
Statistical Analysis 6: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Hazel Nut Wheal; Test type: Superiority or Other; p = 0.226, Chi-squared
Statistical Analysis 7: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Cashew Wheal; Test type: Superiority or Other; p = 0.024, Chi-squared
Statistical Analysis 8: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Walnut Wheal; Test type: Superiority or Other; p = 0.204, Chi-squared
Statistical Analysis 9: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Almond Wheal; Test type: Superiority or Other; p = 0.194, Chi-squared

7. Secondary Outcome: Number of Participants With Food Specific IgE Greater Than or Equal to 0.35 kU/L
Description: At 60 months of age, participants were assessed for potential allergy to selected food allergens. Participants were considered to have a specific food sensitivity if a blood draw showed specific IgE levels greater than or equal to 0.35 kU/L for selected ingested allergens.
Time Frame: 60 months
Population: Intent-to-treat with data available
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Avoidance Group | Peanut Consumption Group
Number analyzed (Participants) | 321 | 319
Participants
  Peanut IgE: number analyzed (Participants) | 307 | 297
  Peanut IgE | 93 | 88
  Egg IgE: number analyzed (Participants) | 307 | 296
  Egg IgE | 120 | 114
  Milk IgE: number analyzed (Participants) | 307 | 296
  Milk IgE | 99 | 105
  Sesame IgE: number analyzed (Participants) | 307 | 296
  Sesame IgE | 89 | 104
  Brazil nut IgE: number analyzed (Participants) | 306 | 296
  Brazil nut IgE | 45 | 55
  Hazel nut IgE: number analyzed (Participants) | 307 | 296
  Hazel nut IgE | 101 | 116
  Cashew IgE: number analyzed (Participants) | 306 | 295
  Cashew IgE | 61 | 73
  Walnut IgE: number analyzed (Participants) | 306 | 295
  Walnut IgE | 52 | 70
  Almond IgE: number analyzed (Participants) | 307 | 296
  Almond IgE | 62 | 71
Statistical Analysis 1: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Peanut IgE; Test type: Superiority or Other; p = 0.859, Chi-squared
Statistical Analysis 2: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Egg IgE; Test type: Superiority or Other; p = 0.885, Chi-squared
Statistical Analysis 3: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Milk IgE; Test type: Superiority or Other; p = 0.403, Chi-squared
Statistical Analysis 4: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Sesame IgE; Test type: Superiority or Other; p = 0.106, Chi-squared
Statistical Analysis 5: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Brazil Nut IgE; Test type: Superiority or Other; p = 0.202, Chi-squared
Statistical Analysis 6: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Hazel Nut IgE; Test type: Superiority or Other; p = 0.108, Chi-squared
Statistical Analysis 7: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Cashew IgE; Test type: Superiority or Other; p = 0.157, Chi-squared
Statistical Analysis 8: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Walnut IgE; Test type: Superiority or Other; p = 0.040, Chi-squared
Statistical Analysis 9: Comparison: Peanut Avoidance Group vs Peanut Consumption Group; Comparison for Almond IgE; Test type: Superiority or Other; p = 0.262, Chi-squared

ADVERSE EVENTS:
Time Frame: Enrollment through last study visit (up to five years)
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group
Serious Adverse Events (participants affected / at risk) | 55/270 | 47/272 | 15/51 | 14/47
Other Adverse Events (participants affected / at risk) | 268/270 | 271/272 | 51/51 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Stratum - Peanut Avoidance Group (N=270) | Negative Stratum - Peanut Consumption Group (N=272) | Positive Stratum - Peanut Avoidance Group (N=51) | Positive Stratum - Peanut Consumption Group (N=47)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 5 (5) | 0 (0) | 7 (9) | 3 (5)
Food allergy (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eczema infected (Infections and infestations) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 9 (12) | 2 (2) | 2 (3)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 17 (25) | 18 (22) | 6 (7) | 6 (7)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Stratum - Peanut Avoidance Group (N=270) | Negative Stratum - Peanut Consumption Group (N=272) | Positive Stratum - Peanut Avoidance Group (N=51) | Positive Stratum - Peanut Consumption Group (N=47)
Conjunctivitis (Eye disorders) | 70 (85) | 45 (48) | 11 (12) | 8 (8)
Constipation (Gastrointestinal disorders) | 23 (30) | 27 (32) | 4 (5) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 60 (64) | 60 (80) | 12 (14) | 7 (9)
Vomiting (Gastrointestinal disorders) | 62 (76) | 70 (100) | 10 (16) | 9 (9)
Pyrexia (General disorders) | 71 (97) | 87 (110) | 10 (13) | 11 (12)
Food allergy (Immune system disorders) | 125 (299) | 132 (286) | 38 (98) | 29 (95)
Hypersensitivity (Immune system disorders) | 14 (16) | 17 (19) | 4 (5) | 7 (7)
Milk allergy (Immune system disorders) | 31 (59) | 29 (47) | 15 (33) | 9 (21)
Seasonal allergy (Immune system disorders) | 39 (49) | 31 (37) | 8 (9) | 9 (11)
Ear infection (Infections and infestations) | 84 (142) | 89 (136) | 10 (15) | 11 (22)
Eczema infected (Infections and infestations) | 41 (55) | 20 (31) | 5 (6) | 8 (14)
Gastroenteritis (Infections and infestations) | 139 (227) | 173 (308) | 29 (44) | 27 (37)
Impetigo (Infections and infestations) | 15 (26) | 17 (21) | 3 (7) | 3 (5)
Lower respiratory tract infection (Infections and infestations) | 98 (164) | 83 (134) | 19 (32) | 20 (30)
Nasopharyngitis (Infections and infestations) | 74 (91) | 86 (112) | 15 (16) | 15 (20)
Otitis media (Infections and infestations) | 34 (42) | 24 (27) | 5 (5) | 7 (7)
Respiratory tract infection (Infections and infestations) | 20 (21) | 22 (24) | 4 (6) | 7 (8)
Rhinitis (Infections and infestations) | 146 (164) | 144 (166) | 38 (42) | 33 (38)
Tonsillitis (Infections and infestations) | 46 (67) | 53 (79) | 8 (11) | 8 (19)
Upper respiratory tract infection (Infections and infestations) | 160 (282) | 191 (399) | 26 (53) | 31 (71)
Varicella (Infections and infestations) | 119 (121) | 145 (153) | 23 (24) | 17 (17)
Viral infection (Infections and infestations) | 44 (48) | 56 (67) | 6 (8) | 10 (14)
Viral upper respiratory tract infection (Infections and infestations) | 30 (34) | 33 (38) | 4 (5) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 60 (81) | 68 (121) | 16 (25) | 17 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (70) | 52 (61) | 8 (13) | 11 (16)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 65 (111) | 58 (111) | 18 (44) | 15 (33)
Eczema (Skin and subcutaneous tissue disorders) | 141 (248) | 147 (243) | 21 (45) | 27 (57)
Rash (Skin and subcutaneous tissue disorders) | 39 (48) | 34 (41) | 6 (6) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 31 (54) | 54 (78) | 9 (12) | 17 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No